CLINICAL TRIAL: NCT03909425
Title: Defining Disease Activity in Neovascular Age-related Macular Degeneration With Optical Coherence Tomography Angiography - A Prospective, Imaging Study - The DANA Study
Brief Title: Defining Disease Activity in Neovascular AMD With Optical Coherence Tomography Angiography
Acronym: DANA
Status: Completed | Type: Observational
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: PATP1032
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: nAMD; Treat and Extend; Aflibercept; OCTA; Neovascular age-related macular degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to be able to describe optical coherence angiography (OCTA) patterns of disease activity and quiescence in eyes that have received treatment. The target population group is patients that have neovascular age-related macular degeneration and have had treatment with aflibercept for this condition.

This is a single-site study and does not involve any masking or treatment allocation.

DETAILED DESCRIPTION:
Treatment of this condition (neovascular age-related macular degeneration - nAMD) with aflibercept has transformed the outlook for patients with this sight-threatening disease.

In clinical practice, eye doctors commonly use a "treat and extend" approach to treatment in which the interval between aflibercept injections is gradually increased once there is nAMD disease quiescence.

It is uncertain about the ideal retinal imaging biomarkers doctors should use to define disease remission or inactivity; and therefore extend treatment intervals. Increased certainty of the ideal biomarker would also avoid stopping treatment too soon.

The scan the investigators will be performing (OCTA imaging) detects blood flow within the choroidal neovascular membrane (CNV) - the immature blood vessel network which causes nAMD. This scan is therefore a potentially powerful way of determining if the disease is active or quiescent. Disease activity on this device can be defined as a blood flow pattern which suggests an active CNV or lesion growth.

By better defining disease activity using OCTA, eye doctors would be more confident in continuing and defining a treatment plan for nAMD.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 50 years of age with a diagnosis of nAMD receiving anti-VEGF treatment with no signs of intra-or subretinal fluid on structural OCT imaging and with no macular haemorrhage after a minimum of three intravitreal injections
* Visual acuity in the study eye of 35 Early Treatment of Diabetic Retinopathy Study (ETDRS) letter score or better (6/60 or better)
* Ability to understand the nature/purpose of the study and to provide informed consent
* Any ocular condition which would lead to image artefact or poor OCT image quality
* Ability to undergo retinal imaging

Exclusion Criteria:

* Patients with polypoidal choroidal vasculopathy or pachychoroid
* Patients in whom imaging of the study eye leads to ungradable OCTA images.
* Any condition which, in the investigators' opinion, would conflict or otherwise prevent the subject from complying with the required procedures, schedule or other study conduct.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with nAMD attending Moorfields Eye Hospital who show no signs of disease activity after treatment with anti-VEGF injections (no signs of macular fluid or macular haemorrhage).
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
Number of participants treated nAMD | 18 Months
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0, Change From Baseline in Pain Scores on the Visual Analog Scale at 6 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Praveen J Patel, FRCOphth, MD, Principal Investigator — Moorfields Eye Hosptial NHS Foundation Trust
Locations (1):
- Moorfields Eye Hospital NHS Foundation Trust, 162 City Road, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No